CLINICAL TRIAL: NCT00513162
Title: Valproate (Valproic Acid) and Etoposide for Patients With Progressive, Relapsed or Refractory Neuronal Tumors and Brain Metastases
Brief Title: Valproate and Etoposide for Patients With Neuronal Tumors and Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0370
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Neuroectodermal Tumor; Brain Metastases; Advanced Cancer
Keywords: Advanced Cancers; Brain; CNS; Neural; Pediatrics; Spinal; Neuroectodermal Tumor; Brain Metastases; Valproate; Valproic Acid; Depakene; Etoposide; VePesid
MeSH Terms: conditions — Neuroectodermal Tumors; Brain Neoplasms | interventions — Valproic Acid; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valproate + Etoposide (Experimental): Valproate Starting Dose of 10 mg/kg By Mouth Daily. Etoposide 25 - 50 mg/m^2 By Mouth Daily.
  Interventions: Drug: Valproate; Drug: Etoposide

INTERVENTIONS:
Drug: Valproate — Starting Dose of 10 mg/kg By Mouth Daily
  Other Names: Valproic Acid; Depakene
Drug: Etoposide — 25 - 50 mg/m^2 By Mouth Daily
  Other Names: VePesid

SUMMARY:
Primary Objective:

* Determine the interindividual range and median of individual maximum tolerated doses of valproic acid administered as one time evening dose in conjunction with a dose oral etoposide (50 mg/m2/day for children, but only 25mg/m2/day for adults to start) for four different age groups.

Secondary Objectives:

* Determine the qualitative and quantitative toxicity and reversibility of toxicity of valproic acid in conjunction with oral etoposide,
* To investigate the clinical pharmacokinetics of valproic acid when given in conjunction with oral etoposide,
* To describe quality of life of patients with relapsed, or progressive central and peripheral nervous system tumors when treated with oral valproic acid and etoposide,
* To observe and describe the response pattern of progressive central nervous system tumors treated with oral valproic acid and etoposide,
* To observe and describe event free survival time and overall survival time of patients with relapsed, or progressive central nervous system tumors when treated with oral valproic acid and etoposide,
* To determine if histone deacetylase activity and topoisomerase expression in lymphocytes of patients is related to valproic acid levels, and
* To determine, if the individual maximal tolerated dose (iMTD) depends on the initial performance status of the patient in the beginning of the treatment.

DETAILED DESCRIPTION:
Study Drugs:

Etoposide is designed to block cell growth by breaking the DNA, which may cause the cells to die.

Valproic acid was first designed as an anti-seizure medication. It was also found to change cancer cells and make them more sensitive to etoposide.

Screening Tests:

Before you start treatment on this study, you will have "screening tests". These tests help your doctor decide if you are eligible to take part in this study.

* Your medical history will be reviewed.
* You will have a physical exam.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation).
* You will complete a questionnaire about your activities or daily living. The questionnaire will take about 5 to 10 minutes to complete.
* Blood (about 2-3 tablespoons) will be drawn for routine tests. This routine blood draw may include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative.
* Urine may be collected to check for metabolic disease. This urine sample may include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative.
* You will have a magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* If your doctor thinks it is necessary, you may have additional blood and/or urine tests.

Dose Escalation:

When you begin the study, you will begin receiving the lowest dose level of valproic acid. Every week, the dose will be increased. This will continue until the maximum tolerated dose (MTD) is found. Once the MTD is found, you will continue to receive that dose level of valproic acid while you are on study. However, if your doctor thinks it is necessary, this dose level could be lowered.

If you are a child (less than or equal to 18 years of age), the amount of etoposide that you take while on study will not change.

If you are an adult (more than 18 years of age), your will receive a low dose of etoposide while the MTD of valproic acid is being found. After the MTD of valproic acid is found, your dose of etoposide will be increased every week until the MTD is found. However, if your doctor thinks it is necessary, this dose level could be lowered.

Study Drug Administration:

You will receive valproic acid and etoposide every evening in pill form.

If you have difficulty swallowing the pills, etoposide can be given in the evening in liquid form. Valproic acid can be given in liquid form, divided in 2 doses per day, 1 in the morning and 1 in the evening.

Study Visits During Dose Escalation:

While your valproic acid or etoposide medication is being increased, every week you will have a physical exam and blood (about 2-3 tablespoons)and urine will be collected for routine tests.

Every other month, you will have CT or MRI scans to check the status of the disease. You may have these tests and procedures more often if your doctor thinks it is necessary.

Study Visits After Maximum Tolerated Dose (MTD):

Every month, you will have a physical exam, and blood (about 2-3 tablespoons) and urine will be collected for routine tests.

Every other month, you will have CT or MRI scans to check the status of the disease.

Every 6 months, a portion of the blood or urine collected for routine tests will be used for a pregnancy test for women who are able to have children.

-You may have these tests and procedures more often if your doctor thinks it is necessary.

Length of Study:

You may remain on study for up to 2 years. You will be taken off study if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

Once you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.
* If your doctor thinks it is necessary, you will have a CT or MRI to check the status of the disease.

Follow-Up:

Once you are off study, you will be contacted by telephone once a year to check the status of the disease. The phone call will take 2-3 minutes.

This is an investigational study. Etoposide is FDA approved and commercially available. Valproic acid is FDA approved and commercially available for the treatment of seizures. The use of these drugs together is investigational. Up to 120 patients will take part in this multicenter study. Up to 100 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diseases: Diagnosis of a neuroectodermal tumor of the central or peripheral nervous system or a brain metastasis.
2. Disease confirmation: Patients must have a diagnosis of a malignant tumor proven by the diagnostic method considered standard of care for the specific tumor.
3. Disease progression and treatment failure: Patient must have failed standard front-line treatment and must not be eligible for any higher-priority therapy.
4. Negative pregnancy test for female patients between menarche and menopause is required.
5. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.
6. Approval for the use of this treatment regimen by the individual's Human Rights Committee or Institutional Review Board (IRB) must be obtained in accordance with the individual institutional policies and the local, state, and national rules, regulations and laws, is mandatory for an enrolling institution. The documentation of this approval must be on file at the MDAnderson Cancer Center Pediatric Oncology Trials Office prior to enrollment of any patient on study.

Exclusion Criteria:

1. Neurofibromatosis type I.
2. Known or suspected inborn errors of metabolism.
3. Patients who require any of the following medications are excluded from enrollment: Carbamazepine, Oxcarbazepine, Primidone, Phenobarbital, Topiramate, Carbapenem antibiotics (ertapenem, imipenem, meropenem), Felbamate, Isoniazid, Lamotrigine, Macrolide antibiotics (clarithromycin, erythromycin, troleandomycin, azithromycin), Zidovudine, Risperidone, Salicylates.
4. Patients who take antiviral medications usually targeted to treat HIV infections or have clinical signs for acquired immunodeficiency syndrome (AIDS) are excluded. HIV testing is not mandatory.
5. Patients who had previous chemotherapy less than three weeks (21 days) ago cannot be enrolled: Patients must have been off all previous chemotherapy or radiotherapy for the 3 weeks prior to initiation of study treatment and recovered from toxic effects of that therapy.
6. Patients which are on a stable dose for valproic acid prior to enrolment are not eligible.
7. Patients which have been treated with valproic acid or other histone deacetylase inhibitors such as SAHAa or MS275 and the treatment has failed to control the tumor are not eligible.
8. Patient which have been treated with oral continuous etoposide previously and the treatment has failed to control the tumor are not eligible.
9. White blood cell count below 2,000/µL excludes patient from enrollment.
10. Absolute neutrophil count below 700/uL excludes patient from enrollment.
11. Platelet count below 80,000 excludes patient from enrollment.
12. Pancreatitis with amylase above two times the upper normal limit excludes patient from enrollment, (even in the absence of clinical signs of pancreatitis).
13. Somnolence at daytime for more than 6 hours excludes patient from enrollment
14. Bilirubin total > 1.5 mg/dL excludes patient from enrollment.
15. ALT > 2.5 times upper normal value excludes patient from enrollment.
16. AST >2.5 x upper normal value excludes patients from enrollment.
17. Frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction) excludes patient from enrollment.
18. Pregnant or nursing women cannot be enrolled.
19. Women of childbearing potential who are not using an effective method of contraception cannot be enrolled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Individual Maximal Tolerated Doses (iMTD) | Continuous assessment and determination of dose-limiting toxicities with each dose level (increasing dose weekly)

CONTACTS AND LOCATIONS:
Overall Officials: Tribhawan S Vats, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org